CLINICAL TRIAL: NCT02607358
Title: NATIS: Non-responders to Antiplatelet Treatment in Acute Ischaemic Stroke
Brief Title: Non-responders to Antiplatelet Treatment in Acute Ischaemic Stroke)
Acronym: NATIS
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-390
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Clopidogrel; acetacylic acid; antiplatelet therapy; HOTPR; VerifyNow
MeSH Terms: conditions — Ischemic Stroke | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Clopidogrel: Clopidogrel non-responders (HOTPR) Blood sampling for HOTPR-testing
  Interventions: Other: blood sampling for HOTPR-testing
- Acetacylicacid: Acetcylicacid non-responders (HOTPR), Blood sampling for HOTPR-testing
  Interventions: Other: blood sampling for HOTPR-testing

INTERVENTIONS:
Other: blood sampling for HOTPR-testing — All subjects are tested for responderstatus using the VerifyNow System

SUMMARY:
Determination of frequency of Clopidigrel- and Acetacylicacid-non-responders (HOTPR) in acute ischemic stroke patients.

DETAILED DESCRIPTION:
Determination of frequency of Clopidigrel- and Acetacylicacid-non-responders (HOTPR) in acute ischemic stroke patients using the VerifyNow system.

ELIGIBILITY:
Inclusion Criteria:

* Suspected acute ischemic stroke and loading dose of Clopidogrel or Acetacylicacid

Exclusion Criteria:

* Previous treatment with platelet inhibitor
* NOAC or Vitamin K-antagonist treatment
* Final diagnosis other than Ischemoc stroke or Transitoric ischemic attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Ischemic stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Responder status | immediately
  Platelet reactivity with PRU measurement

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Rath, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Neurologisk afdeling, Roskilde, Denmark